CLINICAL TRIAL: NCT02467595
Title: The Effect of no Muscle Relaxant Versus Reduced-dose Rocuronium on the Anesthetic Condition With Fentanyl in Children Undergoing Adenotonsillectomy
Brief Title: The Effect of no Muscle Relaxant Versus Reduced-dose Rocuronium on Anesthesia in Adenotonsillectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Sangjae Park, Resident, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ED14142
Record Dates: First submitted 2015-05-11; First posted 2015-06-10 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Muscle Relaxants
Keywords: no muscle relaxant; rocuronium; intubation condition; tracheal intubation; operating room time; low-dose rocuronium
MeSH Terms: conditions — Muscle Hypotonia | interventions — Rocuronium; Fentanyl; Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- R 0.15 group (Experimental): Rocuronium bromide 0.15 mg kg-1 group
  1. Anesthesia was induced with propofol 2.5 mg kg-1 , fentanyl 2 mcg kg-1, and rocuronium bromide 0.15 mg kg-1
  2. After mask ventilation with 5 vol% sevoflurane in 100% oxygen for 2 minutes, tracheal intubation was done.
  3. At the end of surgery, discontinuation of sevoflurane and extubation, sending recovery room.
  4. When poor intubating condition., added rocuronium bromide 0.3 mg kg-1 .
  Drug: Rocuronium bromide Rocuronium bromide 0.15 mg kg-1 was injected at I.V. line to patients (R 0.15 group), as muscle relaxants during anesthesia for adenotonsillectomy.
  Interventions: Drug: Rocuronium bromide 0.15 mg kg-1; Drug: Fentanyl; Drug: Propofol; Drug: Sevoflurane
- R 0.3 group (Active Comparator): Rocuronium bromide 0.3 mg kg-1 group
  1. Anesthesia was induced with propofol 2.5 mg kg-1 , fentanyl 2 mcg kg-1, and rocuronium bromide 0.3 mg kg-1
  2. After mask ventilation with 5 vol% sevoflurane in 100% oxygen for 2 minutes, tracheal intubation was done.
  3. At the end of surgery, discontinuation of sevoflurane and extubation, sending recovery room.
  4. When poor intubating condition., added rocuronium bromide 0.3 mg kg-1 .
  Drug: Rocuronium bromide Rocuronium bromide 0.3 mg kg-1 was injected at I.V. line to patients (R 0.3 group), as muscle relaxants during anesthesia for adenotonsillectomy.
  Interventions: Drug: Rocuronium bromide 0.3 mg kg-1; Drug: Fentanyl; Drug: Propofol; Drug: Sevoflurane
- S group (Placebo Comparator): saline
  1. Anesthesia was induced with propofol 2.5 mg kg-1 , fentanyl 2 mcg kg-1, and saline.
  2. After mask ventilation with 5 vol% sevoflurane in 100% oxygen for 2 minutes, tracheal intubation was done.
  3. At the end of surgery, discontinuation of sevoflurane and extubation, sending recovery room.
  4. When poor intubating condition., added rocuronium bromide0.3 mg kg-1 .
  Interventions: Drug: Fentanyl; Drug: Propofol; Drug: Sevoflurane

INTERVENTIONS:
Drug: Rocuronium bromide 0.15 mg kg-1 — Rocuronium bromide 0.15 mg kg-1 was injected at I.V. line to patients (R 0.15 group), as muscle relaxants during anesthesia for adenotonsillectomy.
  Other Names: Esmerone
  Arms: R 0.15 group
Drug: Rocuronium bromide 0.3 mg kg-1 — Rocuronium 0.3 mg kg-1 was injected at I.V. line to patients (R 0.3 group), as muscle relaxants during anesthesia for adenotonsillectomy.
  Other Names: Esmerone
  Arms: R 0.3 group
Drug: Fentanyl — Fentanyl 2 mcg kg-1 was injected at I.V. line to patients
  Other Names: 하나구연산펜타닐주사
Drug: Propofol — Propofol 2.5 mg kg-1 was injected at I.V. line to patients
  Other Names: Fresofol MCT 1%
Drug: Sevoflurane — After mask ventilation with 5 vol% sevoflurane in 100% oxygen for 2 minutes, tracheal intubation was done.
  Other Names: 세보프란 흡입액

SUMMARY:
This study aimed to compare the effect of no muscle relaxants and reduced-dose rocuronium on the anesthetic induction and emergence with fentanyl in children undergoing adenotonsillectomy.

DETAILED DESCRIPTION:
Adenotonsillectomy in children is a short surgical procedure under general anesthesia. The ideal muscle relaxant requires intense neuromuscular block for optimal surgical work and complete recovery of neuromuscular function immediately after the end of the surgical procedure without postoperative morbidity. Rocuronium is an intermediate acting neuromuscular blockade. Reduced-dose rocuronium has been reported to provide optimal anesthetic induction without delayed recovery. The investigators aimed to compare the effect of no muscle relaxants and reduced-dose rocuronium on the anesthetic induction and emergence with fentanyl in children undergoing adenotonsillectomy.

After Institutional Review Board approval and written informed consent from the parents were obtained, 75 children (aged 3 to 10 years, ASA(The American Society of Anesthesia ) I or II) scheduled for adenotonsillectomy were included. Anesthesia was induced with propofol 2.5 mg kg-1 , fentanyl 2 mcg kg-1, and rocuronium 0.15 mg kg-1 (R 0.15 group) or rocuronium 0.3mg kg-1 (R 0.3 group) or saline (S group). After mask ventilation with 5 vol% sevoflurane in 100% oxygen for 2 minutes, tracheal intubation was done. The investigators assessed conditions during tracheal intubation as excellent, good or poor, using five variables; jaw relaxation, vocal cord position, vocal cord movement, coughing, and movement of the limbs. The investigators added rocuronium 0.3 mg kg-1 when there was more than one poor condition. The investigators recorded the time from discontinuation of sevoflurane to time to extubation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist[ASA] class 1-2
* scheduled adenotonsillectomy
* written informed consent

Exclusion Criteria:

* allergy of opioids, neuromuscular blocking drugs or other medications used during general anesthesia
* known or suspected upper respiratory infection
* disorder affecting neuromuscular blockade
* suspected difficult tracheal intubation
* Developmental Disability
* known or suspected psychologic disorder
* medication (psychoactive drugs)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Conditions during tracheal intubation | At the time to tracheal intubation, after mask ventilation for 2 minutes
  We assessed conditions during tracheal intubation as excellent, good or poor, and additionally using five variables; jaw relaxation, vocal cord position, vocal cord movement, coughing, and movement of the limbs.

SECONDARY OUTCOMES:
time to extubation | intraoperatve
  When surgery is end, we discontinue sevoflurane for maintaining anesthesia. So we check the time of this point until extubation.

OTHER OUTCOMES:
Additive rocuronium | intraoperatve
  We added rocuronium 0.3 mg kg-1 when there was more than one poor intubating condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jang Eun Cho, M.D.,Ph.D., Principal Investigator — Anesthesia and pain medicine department, Korea University Anam Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huh H, Park JJ, Kim JY, Kim TH, Yoon SZ, Shin HW, Lee HW, Lim HJ, Cho JE. Optimal dose of rocuronium bromide undergoing adenotonsillectomy under 5% sevoflurane with fentanyl. Int J Pediatr Otorhinolaryngol. 2017 Oct;101:70-74. doi: 10.1016/j.ijporl.2017.07.030. Epub 2017 Jul 25. PMID 28964314